CLINICAL TRIAL: NCT02258399
Title: Exercise in the Fasted State, Glucose Metabolism and Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: University of Stirling (Other); University of Birmingham (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Lecturer, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RE-FH1109
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Energy Balance; Blood Glucose
MeSH Terms: interventions — Exercise; Breakfast

ARMS (3):
- Breakfast Rest (Active Comparator)
  Interventions: Dietary Supplement: Breakfast
- Breakfast Exercise (Active Comparator)
  Interventions: Behavioral: Exercise; Dietary Supplement: Breakfast
- Fasted Exercise (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Moderate intensity exercise
  Arms: Breakfast Exercise; Fasted Exercise
Dietary Supplement: Breakfast — Breakfast consumption
  Arms: Breakfast Exercise; Breakfast Rest

SUMMARY:
The ability to control our blood glucose (sugar) concentrations after a meal is a strong predictor of the risk of disease. Our bodies respond to glucose ingestion by reducing the amount of glucose from the liver entering the bloodstream. At the same time muscle increases the amount of glucose it take up from the bloodstream. This ensures that our blood glucose levels do not get too high. The investigators want to understand what happens to these processes following exercise after breakfast and after an overnight fast. In addition, the investigators also want to understand whether exercising with or without breakfast influences our appetite, food intake and activity levels later in the day.

ELIGIBILITY:
Inclusion Criteria:

* Males.
* Aged 18-49.
* Individuals free from known cardiovascular, metabolic or joint disease as determined by standard health questionnaire.
* Habitual regularly participating in exercise (minimum of 3 sessions per week on average)
* Non-smoker

Exclusion Criteria:

* Known or suspected food intolerances, allergies or hypersensitivity.
* Any bleeding disorder or taking medication which impacts blood coagulation.
* Known tendency towards keloid scarring.
* Known sensitivity or allergy to any local anaesthetic medicines.
* Any reported use of substances which may pose undue personal risk to participants or introduce bias into the experiment.
* Any other condition or behaviour deemed either to pose undue personal risk to participants or introduce bias into the experiment.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Exogenous glucose appearance rate | 120 minutes
  Exogenous glucose appearance rates following an oral glucose tolerance test (total appearance over 120 minutes).
Energy balance | 24 hours
  Energy balance (intake minus expenditure) over 24 h from the beginning of the trial

SECONDARY OUTCOMES:
Endogenous glucose appearance rates | 120 minutes
  Endogenous glucose appearance rates following an oral glucose tolerance test (total appearance over 120 minutes).
Glucose clearance rates | 120 minutes
  Glucose clearance rates following an oral glucose tolerance test (total clearance over 120 minutes).
Energy intake | 24 h
  Weighted energy intake over 24 hours from the beginning of the trial.
Energy expenditure | 24 h
  Energy expenditure, derived from indirect calorimetry, acccelerometry and heart rate monitoring.
Exogenous glucose appearance rates | 120 minutes
  Exogenous glucose appearance rates following an oral glucose tolerance test (total appearance over 120 minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom

REFERENCES:
- [Background] Gonzalez JT. Paradoxical second-meal phenomenon in the acute postexercise period. Nutrition. 2014 Sep;30(9):961-7. doi: 10.1016/j.nut.2013.12.001. Epub 2013 Dec 14. PMID 24986552
- [Background] Gonzalez JT, Veasey RC, Rumbold PL, Stevenson EJ. Breakfast and exercise contingently affect postprandial metabolism and energy balance in physically active males. Br J Nutr. 2013 Aug;110(4):721-32. doi: 10.1017/S0007114512005582. Epub 2013 Jan 29. PMID 23340006
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Edinburgh RM, Hengist A, Smith HA, Travers RL, Betts JA, Thompson D, Walhin JP, Wallis GA, Hamilton DL, Stevenson EJ, Tipton KD, Gonzalez JT. Skipping Breakfast Before Exercise Creates a More Negative 24-hour Energy Balance: A Randomized Controlled Trial in Healthy Physically Active Young Men. J Nutr. 2019 Aug 1;149(8):1326-1334. doi: 10.1093/jn/nxz018. PMID 31321428